CLINICAL TRIAL: NCT05190523
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of ASC42 Tablets in Subjects With Primary Biliary Cholangitis
Brief Title: Study to Evaluate the Safety and Efficacy of ASC42 Tablets in Subjects With Primary Biliary Cholangitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gannex Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC42-202
Record Dates: First submitted 2021-12-13; First posted 2022-01-13 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Primary Biliary Cholangitis
Keywords: ASC42; primary biliary cholangitis; PBC
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ASC42 tablets of 5mg (Experimental): ASC42 tablets 5mg for 12 weeks
  Interventions: Drug: ASC42 5 mg
- ASC42 tablets of 10mg (Experimental): ASC42 tablets 10mg for 12 weeks
  Interventions: Drug: ASC42 10 mg
- ASC42 tablets of 15mg (Experimental): ASC42 tablets 15mg for 12 weeks
  Interventions: Drug: ASC42 15 mg
- Placebo (Placebo Comparator): Placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASC42 5 mg — 5 mg of ASC42 tablets orally once daily for 12 weeks.
  Arms: ASC42 tablets of 5mg
Drug: ASC42 10 mg — 2 x 5 mg of ASC42 tablets orally once daily for 12 weeks.
  Arms: ASC42 tablets of 10mg
Drug: ASC42 15 mg — 15 mg of ASC42 tablets orally once daily for 12 weeks.
  Arms: ASC42 tablets of 15mg
Drug: Placebo — Placebo tablets orally once daily for 12 weeks.
  Arms: Placebo

SUMMARY:
This study is a phase II, multicenter, randomized, double-blind, placebo-controlled, seamless adaptive design clinical study, aiming to evaluate the safety and effectiveness of three doses of ASC42 matched placebo in subjects with primary biliary cholangitis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤75 years old at screening.
* Definite or probable PBC diagnosis, as demonstrated by the presence of ≥ 2 of the following 3 diagnostic factors:

  1. Biochemical evidence of cholestasis based on ALP elevation.
  2. Presence of AMA, or other PBC-specific autoantibodies, including sp100 or gp210, if AMA is negative.
  3. Liver biopsy consistent with PBC.
* Screening ALP ≥ 1.67× ULN
* Taking UDCA for at least 6 months (stable dose for ≥ 3 months) prior to Day 0, or unable to tolerate UDCA (no UDCA for ≥ 3 months) prior to Day 0.

Exclusion Criteria:

* ALT or AST > 5× ULN; ALP >10× ULN
* History or presence of other concomitant liver diseases
* Child-Pugh grade B or C

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Percentage changes of alkaline phosphatase (ALP) compared with baseline. | Day85

SECONDARY OUTCOMES:
Percentage changes and absolute changes of alkaline phosphatase (ALP) compared with baseline. | Day15\29\57\85
Percentage changes and absolute changes of serum γ-glutamyltransferase (GGT), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) compared with baseline. | Day15\29\57\85
Incidence of treatment-emergent adverse events, serious adverse events and adverse events of special interests. | Day15\29\57\85

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China